CLINICAL TRIAL: NCT01536717
Title: Comparison of Periosteal and Subcutaneous Infusions of Articaine and Bupivacaine in Treatment of Acute Pain After Sternotomy
Brief Title: Comparison of the Local Anaesthetics Articaine and Bupivacaine in Treatment of Acute Sternum Pain After Heart Surgery
Status: Suspended | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Reino Poyhia, MD, PhD, Docent, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011-004307-20
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Diseases of Mitral Valve; Aortic Valve Disorder; Atrial Septal Defects; Intracardiac Myxoma
Keywords: atrial septal defect; mitral valve annuloplasty; aortic valve annuloplasty; open heart surgery; oxycodone consumption; articain; bupivacaine; pain after sternotomy; postoperative pain; wound infusion
MeSH Terms: conditions — Aortic Valve Disease; Heart Septal Defects, Atrial; Atrial myxoma, familial; Pain, Postoperative | interventions — Carticaine; Solutions; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine hydrochloride 0.5% (Active Comparator): Bupivacaine hydrochloride is related chemically and pharmacologically to the aminoacyl local anesthetics. Bupivacaine hydrochloride is indicated for the production of local or regional anesthesia or analgesia for surgery, for oral surgery procedures, for diagnostic and therapeutic procedures, and for obstetrical procedures.
  Interventions: Drug: Articaine hydrochloride 2% solution
- Sodium chloride 0,9% (Placebo Comparator)
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: Articaine hydrochloride 2% solution — * 4 ml/h periosteal wound infusion
  * duration of 72 h
  Other Names: Ultracain D ohne Adrenalin 20 mg/ml, ATC code N01BB08
  Arms: Bupivacaine hydrochloride 0.5%
Drug: Sodium Chloride — Placebo Sodium chloride 0,9%
  Arms: Sodium chloride 0,9%

SUMMARY:
The purpose of this study is to examine the wound infusion of articaine for treatment of acute post-sternotomy pain in a placebo-controlled manner using a prospective and randomized design and an active control (bupivacaine)

DETAILED DESCRIPTION:
Acute pain after open heart surgery can be moderate or strong and is mostly caused by sternotomy. Pain is the worst during the first two post-operative days and, if not adequately treated, can delay the patient´s recovery from surgery. Sternotomy pain can be alleviated by using paracetamol, non-steroidal anti-inflammatory drugs (NSAIDs) and opioids. All these drugs may have remarkable side-effects which may delay the recovery from surgery: opioids are respiratory depressants and slower the gastrointestinal motility, NSAIDs reduce intrarenal blood flow and may disturb coagulation. Post-operative opioid consumption can be reduced by using wound infiltration analgesia.

The use of wound infiltration analgesia has not been extensively investigated in treatment of acute pain after sternotomy. There is some evidence, that 0.5% bupivacaine reduces the acute post-sternotomy pain when infused constantly via catheters placed under the fascia (periosteal placement) and the skin.

During 48 hours infusion toxic bupivacaine plasma levels were not observed. There is an evidence that local anesthetics can be bacteriostatic both in vitro and in vivo.

Articaine is an amide-type local anesthetics, which has been used extensively in dental procedures since more than forty years. It has been successfully used in infiltration, epidural, spinal and other regional anesthesia procedures. Articaine is quickly hydrolyzed in plasma and excreted by kidneys. Clearance of articain (500-1110l/h) is faster than that of lidocaine (68l/h) and it is also the reason for articaine´s low toxicity profile. Because of it´s low toxicity and high ability to penetrate the periosteal tissue, articaine may be advantageous in treatment of acute pain after sternotomy, but aforementioned indication for use of articaine has not been investigated. Compared to other local anesthetics, articaine in high concentration has the same neurotoxicity profile, when injected directly into rat´s sciatic nerve. Articaine has not been extensively compared to other local anesthetics, but according the latest odontologic investigation, single dose 0.5% bupivacaine and single-dose 4% articaine were comparable in their analgesic effects during tooth extraction procedure. There are no controlled randomized trials comparing analgesic effect of articaine and other local anesthetics infusions.

In our investigation bupivacain 0.5 % was chosen as an active control, because it has appeared effective in acute postoperative pain and it has reduced the need for opioid analgetics after sternotomy

ELIGIBILITY:
Inclusion Criteria:

* elective procedure
* open heart surgery
* aortic valve surgery
* mitral valve surgery
* atrial septal defect repair surgery
* intracardial myxoma removal surgery

Exclusion Criteria:

* local anesthetic allergy
* sulphide allergy
* asthma
* pregnant women
* neurological disease (TIA excluded)
* congestive heart failure
* left ventricle ejection fracture under 0.3
* liver failure
* diabetes mellitus with documented polyneuropathy
* chronic pain condition
* mother tongue not finnish or swedish
* patients, who do not agree blood transfusions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-03; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Oxycodone consumption | 72 hours from initiation of treatment

SECONDARY OUTCOMES:
Intensity of pain in rest/in movement (AUC) | 72 hours from initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Reino Pöyhiä, MD, PhD, Study Chair — Department of Anesthesiology and Intensive care, Division of Surgery, Meilahti Hospital, Helsinki University Central Hospital; Mihkel Meinberg, MD, Principal Investigator — Department of Anesthesiology and Intensive care medicine, Division of Surgery, Meilahti Hospital, Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Department of Anesthesiology and Intensive care medicine, Divison of Surgery, Meilahti hospital, Helsinki University Central Hospital, Helsinki, Uusimaa
  - Department of Cardiothoracic surgery, Division of Surgery, Meilahti hospital, Helsinki University Central Hospital, Helsinki, Uusimaa

REFERENCES:
- [Background] Kehlet H, Andersen LO. Local infiltration analgesia in joint replacement: the evidence and recommendations for clinical practice. Acta Anaesthesiol Scand. 2011 Aug;55(7):778-84. doi: 10.1111/j.1399-6576.2011.02429.x. Epub 2011 Apr 4. PMID 21463261
- [Background] White PF, Rawal S, Latham P, Markowitz S, Issioui T, Chi L, Dellaria S, Shi C, Morse L, Ing C. Use of a continuous local anesthetic infusion for pain management after median sternotomy. Anesthesiology. 2003 Oct;99(4):918-23. doi: 10.1097/00000542-200310000-00026. PMID 14508326
- [Background] Magnano D, Montalbano R, Lamarra M, Ferri F, Lorini L, Clarizia S, Rescigno G. Ineffectiveness of local wound anesthesia to reduce postoperative pain after median sternotomy. J Card Surg. 2005 Jul-Aug;20(4):314-8. doi: 10.1111/j.1540-8191.2005.200318.x. PMID 15985128
- [Background] Pere P, Lindgren L, Vaara M. Poor antibacterial effect of ropivacaine: comparison with bupivacaine. Anesthesiology. 1999 Sep;91(3):884-6. doi: 10.1097/00000542-199909000-00047. No abstract available. PMID 10485806
- [Background] Vree TB, Gielen MJ. Clinical pharmacology and the use of articaine for local and regional anaesthesia. Best Pract Res Clin Anaesthesiol. 2005 Jun;19(2):293-308. doi: 10.1016/j.bpa.2004.12.006. PMID 15966499
- [Background] Pelz K, Wiedmann-Al-Ahmad M, Bogdan C, Otten JE. Analysis of the antimicrobial activity of local anaesthetics used for dental analgesia. J Med Microbiol. 2008 Jan;57(Pt 1):88-94. doi: 10.1099/jmm.0.47339-0. PMID 18065672
- [Background] Vree TB, Baars AM, van Oss GE, Booij LH. High-performance liquid chromatography and preliminary pharmacokinetics of articaine and its 2-carboxy metabolite in human serum and urine. J Chromatogr. 1988 Feb 26;424(2):440-4. doi: 10.1016/s0378-4347(00)81126-3. No abstract available. PMID 3372637
- [Background] Brinklov MM. Clinical effects of carticaine, a new local anesthetic. A survey and a double-blind investigation comparing carticaine with lidocaine in epidural analgesia. Acta Anaesthesiol Scand. 1977;21(1):5-16. doi: 10.1111/j.1399-6576.1977.tb01186.x. PMID 320810
- [Background] Kallio H, Snall EV, Luode T, Rosenberg PH. Hyperbaric articaine for day-case spinal anaesthesia. Br J Anaesth. 2006 Nov;97(5):704-9. doi: 10.1093/bja/ael222. Epub 2006 Aug 5. PMID 16891634
- [Background] Pitkanen MT, Xu M, Haasio J, Rosenberg PH. Comparison of 0.5% articaine and 0.5% prilocaine in intravenous regional anesthesia of the arm: a cross-over study in volunteers. Reg Anesth Pain Med. 1999 Mar-Apr;24(2):131-5. PMID 10204898
- [Background] Simon MA, Vree TB, Gielen MJ, Booij LH, Lagerwerf AJ. Similar motor block effects with different disposition kinetics between lidocaine and (+ or -) articaine in patients undergoing axillary brachial plexus block during day case surgery. Int J Clin Pharmacol Ther. 1999 Dec;37(12):598-607. PMID 10599952
- [Background] Trullenque-Eriksson A, Guisado-Moya B. Comparative study of two local anesthetics in the surgical extraction of mandibular third molars: bupivacaine and articaine. Med Oral Patol Oral Cir Bucal. 2011 May 1;16(3):e390-6. doi: 10.4317/medoral.16.e390. PMID 21196829
- [Background] Pesonen A, Suojaranta-Ylinen R, Hammaren E, Kontinen VK, Raivio P, Tarkkila P, Rosenberg PH. Pregabalin has an opioid-sparing effect in elderly patients after cardiac surgery: a randomized placebo-controlled trial. Br J Anaesth. 2011 Jun;106(6):873-81. doi: 10.1093/bja/aer083. Epub 2011 Apr 6. PMID 21474474
- [Background] Hillerup S, Bakke M, Larsen JO, Thomsen CE, Gerds TA. Concentration-dependent neurotoxicity of articaine: an electrophysiological and stereological study of the rat sciatic nerve. Anesth Analg. 2011 Jun;112(6):1330-8. doi: 10.1213/ANE.0b013e3182172a2e. Epub 2011 Apr 5. PMID 21467556
- [Background] Tirotta CF, Munro HM, Salvaggio J, Madril D, Felix DE, Rusinowski L, Tyler C, Decampli W, Hannan RL, Burke RP. Continuous incisional infusion of local anesthetic in pediatric patients following open heart surgery. Paediatr Anaesth. 2009 Jun;19(6):571-6. doi: 10.1111/j.1460-9592.2009.03009.x. PMID 19645974
- [Background] Hynninen MS, Cheng DC, Hossain I, Carroll J, Aumbhagavan SS, Yue R, Karski JM. Non-steroidal anti-inflammatory drugs in treatment of postoperative pain after cardiac surgery. Can J Anaesth. 2000 Dec;47(12):1182-7. doi: 10.1007/BF03019866. PMID 11132739
- [Background] Lahtinen P, Kokki H, Hendolin H, Hakala T, Hynynen M. Propacetamol as adjunctive treatment for postoperative pain after cardiac surgery. Anesth Analg. 2002 Oct;95(4):813-9, table of contents. doi: 10.1097/00000539-200210000-00005. PMID 12351250
- [Background] Mueller XM, Tinguely F, Tevaearai HT, Revelly JP, Chiolero R, von Segesser LK. Pain location, distribution, and intensity after cardiac surgery. Chest. 2000 Aug;118(2):391-6. doi: 10.1378/chest.118.2.391. PMID 10936130
- [Background] Oertel R, Rahn R, Kirch W. Clinical pharmacokinetics of articaine. Clin Pharmacokinet. 1997 Dec;33(6):417-25. doi: 10.2165/00003088-199733060-00002. PMID 9435991
- [Background] Simon MA, Vree TB, Gielen MJ, Booij LH. Comparison of the effects and disposition kinetics of articaine and lidocaine in 20 patients undergoing intravenous regional anaesthesia during day case surgery. Pharm World Sci. 1998 Apr;20(2):88-92. doi: 10.1023/a:1008622018161. PMID 9584343